CLINICAL TRIAL: NCT06564610
Title: Laparoscopic Transversus Abdominis Plane Block Versus Erector Spinae Plane Block in Obese Patients Undergoing Bariatric Surgery: a Randomized Controlled Trial
Brief Title: Laparoscopic Transversus Abdominis Plane Block Versus Erector Spinae Plane Block in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD-292-2022
Record Dates: First submitted 2024-08-16; First posted 2024-08-21 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-08

CONDITIONS: Pain, Postoperative; Obesity; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Obesity; Agnosia | interventions — Bariatric Surgery; Intubation, Intratracheal; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transversus abdominis block (Experimental): Patients in this group will receive Transversus Abdominis block guided by the laparoscope at the beginning of surgery.
  Interventions: Procedure: Transversus abdominis block; Procedure: Bariatric surgery; Device: Endotracheal intubation; Drug: Propofol
- Erector spinae block (Active Comparator): Patients in this group will receive Erector Spinae block guided by the ultrasound after induction of anesthesia.
  Interventions: Procedure: Erector spinae block; Procedure: Bariatric surgery; Device: Endotracheal intubation; Drug: Propofol

INTERVENTIONS:
Procedure: Transversus abdominis block — The block will be performed by the surgeon by injecting local anesthetic at the beginning of surgery under the guidance of the laparoscope.
  Arms: Transversus abdominis block
Procedure: Erector spinae block — The block will be performed by the anesthetist by injecting local anesthetic after induction of anesthesia under the guidance of the ultrasound.
  Arms: Erector spinae block
Procedure: Bariatric surgery — Laparoscopic bariatric procedure will be performed
Device: Endotracheal intubation — An endotracheal tube will be inserted as a part of general anesthesia to all patients
Drug: Propofol — The patients will receive propofol for induction of anesthesia

SUMMARY:
The aim of this work is to compare the analgesic efficacy of laparoscopic transversus abdominis plane block, performed by the surgeon to ultrasound-guided erector spinae plane block, performed by the anesthetist, in patients with obesity undergoing bariatric surgery.

DETAILED DESCRIPTION:
This is a randomized controlled trial which will include patients with obesity undergoing bariatric surgery. The patients will be randomly allocated into two groups: transversus abdominis plane block group and erector spinae plane block group. The block will be performed after induction of general anesthesia. Preoperative evaluation and preparation will include history-taking, laboratory investigation, fasting recommendations, and optimization of the medical status. The two groups will receive standard induction and maintenance of anesthesia. After the end of the operation, patients will receive standard care according to the local protocols and the enhanced recovery recommendations. Patients will be monitored according to the pain-related outcomes as well as hemodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with obesity undergoing laparoscopic bariatric surgery under general anesthesia.

Exclusion Criteria:

* Allergy to local anaesthetic.
* Bleeding disorders.
* Obstructive sleep apnea.
* inability to understand the numerical rating scale for pain assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale | 24 hours after surgery
  This is a scale for pain assessment which ranges between 0 and 10 with the highest level of pain having score 10 and lowest level of pain having score 0

SECONDARY OUTCOMES:
Consumption of analgesia | 24 hours after surgery
  This is the total consumption of nalbuphine by the patient measured in milligrams
Heart rate | 24 hours after surgery
  This is the number of heart beats measured as frequency of heart beats in one minute.
Systolic blood pressure | 24 hours after surgery
  This is the systolic arterial blood pressure measured in mmHg.
Vomiting | 24 hours
  This is the incidence of vomiting after surgery measured as the frequency of patients with vomiting.
Diastolic blood pressure | 24 hours
  This is the diastolic arterial blood pressure measured in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hasanin, Professor, Principal Investigator — Professor of anesthesia
Locations (1):
- Faculty of medicine, Cairo University., Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No